CLINICAL TRIAL: NCT01845987
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of CNTO 1959, a Human Anti-IL 23 Monoclonal Antibody, Following Subcutaneous Administration in Subjects With Palmoplantar Pustulosis
Brief Title: A Study of the Efficacy, Safety and Tolerability of CNTO 1959, a Human Anti-IL 23 Monoclonal Antibody in Participants With Palmoplantar Pustulosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100950; CNTO1959PPP2001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Palmoplantaris Pustulosis
Keywords: Palmoplantaris Pustulosis; CNTO 1959; Psoriasis; Anti-IL 23 Monoclonal Antibody
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CNTO 1959 (Experimental)
  Interventions: Drug: CNTO 1959

INTERVENTIONS:
Drug: Placebo — Placebo, as two 1-ml subcutaneous (SC) injections, at Week 0 and Week 4
  Arms: Placebo
Drug: CNTO 1959 — CNTO 1959 200 mg, as two 1-ml subcutaneous (SC) injections, at Week 0 and Week 4
  Arms: CNTO 1959

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of CNTO 1959 following subcutaneous administration in participants with palmoplantar pustulosis.

DETAILED DESCRIPTION:
This will be a double-blind (participants and study personnel will not know the identity of the treatments given), multicenter study that is placebo-controlled (a placebo is identical to a study treatment, but has no active ingredients). Participants will be randomly assigned to 1 of 2 treatment groups (CNTO 1959 or placebo). The total duration of participation will be approximately 30 weeks, including a screening period of about 6 weeks before dosing. Participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of palmoplantar pustulosis at screening (participants with concurrent extra-palmoplantar lesions [includes plaque-type psoriasis lesions] and/or pustulotic arthro-osteitis [PAO] can also be included)
* Participant has active lesions on the palms or soles at screening and baseline
* Participant has inadequate response to treatment with topical steroid and/or topical vitamin D3 derivative preparations and/or phototherapy and/or systemic etretinate prior to or at screening
* Participant has a Palmoplantar Pustulosis Severity Index (PPSI) score of 7 or greater at screening and baseline
* At screening, the results of laboratory blood tests must be within protocol-specified limits

Exclusion Criteria:

* History of or current signs of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurologic, cerebral, or psychiatric disease
* Participant has unstable cardiovascular disease, defined as a recent clinical deterioration in the last 3 months or a cardiac hospitalization within the last 3 months prior to screening
* History of chronic or recurrent infectious disease, including, but not limited to, chronic renal infection, chronic chest infection (eg, bronchiectasis), recurrent urinary tract infection (eg, recurrent pyelonephritis), fungal infection (eg, mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers
* Participant has or has had a serious infection (eg, sepsis, pneumonia or pyelonephritis), or has been hospitalized or received intravenous (IV) antibiotics for an infection during the 2 months prior to screening
* Participant has or has had herpes zoster within the 2 months prior to screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PPSI total score at Week 16. | Baseline to Week 16
  The Palmoplantar Pustulosis Severity Index (PPSI) assesses the severity of palmoplantar pustulosis lesions and their response to therapy. Scores can range from 0 to 12, with higher scores indicating more severity.

SECONDARY OUTCOMES:
Change from baseline in PPSI total score over time | Baseline up to 24 weeks
  The Palmoplantar Pustulosis Severity Index (PPSI) assesses the severity of palmoplantar pustulosis lesions and their response to therapy. Scores can range from 0 to 12, with higher scores indicating more severity.
Change from baseline in PPPASI total score | Baseline up to 24 weeks
  The Palmoplantar Pustulosis Area and Severity Index (PPPASI) assesses the severity of palmoplantar pustulosis lesions and their response to therapy. Scores can range from 0 to 72, with higher scores indicating more severity.
Proportion of participants who achieve a PPPASI-50 | Up to 24 weeks
  PPPASI-50 is at least 50% reduction in the PPPASI score.
Proportion of participants who achieve a PGA score of 1 or less | Up to 24 weeks
  The Physician's Global Assessment (PGA) is used to determine the participant's overall palmoplantar pustulosis lesions, at a given time point. Scores can range from 0 (clear) to 5 (very severe).
Proportion of participants who achieve a PPPASI-75 | Up to 24 weeks
  PPPASI-75 is at least 75% reduction in the PPPASI score.
Change from baseline in PA (each score) | Baseline up to 24 weeks
  The Physician's Assessment (PA) is used to determine the participant's pustule, vesicle, and nail lesions at a given time point. Scores can range from 0 (clear) to 5 (very severe).
Change from baseline in Patient's VAS-PPP severity | Baseline up to 24 weeks
  The Patient's Visual Analogue Scale (VAS) assessment of palmoplantar pustulosis severity will be recorded on a 10-cm VAS.
Change from baseline in Physician's VAS-PAO activity | Baseline up to 24 weeks
  Physician's Visual Analogue Scale Assessment of Pustulotic Arthro-Osteitis Activity will be recorded on a 10-cm VAS.
Change from baseline in Patient's VAS-PAO activity and pain | Baseline up to 24 weeks
  Patient's Visual Analogue Scale Assessment of Pustulotic Arthro-Osteitis Activity and Pain will be recorded on each 10-cm VAS.
Change from baseline in Dermatology Life Quality Index (DLQI) | Baseline up to 24 weeks
  The DLQI is a 10-item questionnaire that in addition to evaluating overall quality of life (QOL), can be used to assess 6 different aspects that may affect QOL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment.
Change form baseline in SF-36 score | Baseline up to 24 weeks
  The 36-Item Short Form Health Survey (SF-36) consists of 8 multi-item scales: limitations in physical functioning due to health problems, limitations in usual role activities due to physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities due to personal or emotional problems, limitations in social functioning due to physical or mental health problems, vitality (energy and fatigue), and general health perception.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (8):
- Japan (8):
  - Asahikawa
  - Fukuoka
  - Fukushima
  - Matsumoto
  - Sapporo
  - Sendai
  - Tokyo
  - Touon

REFERENCES:
- [Derived] Terui T, Kobayashi S, Okubo Y, Murakami M, Hirose K, Kubo H. Efficacy and Safety of Guselkumab, an Anti-interleukin 23 Monoclonal Antibody, for Palmoplantar Pustulosis: A Randomized Clinical Trial. JAMA Dermatol. 2018 Mar 1;154(3):309-316. doi: 10.1001/jamadermatol.2017.5937. PMID 29417135